CLINICAL TRIAL: NCT01672853
Title: A Phase 2b, Dose-Ranging, Randomized, Double-Blind, Placebo-Controlled Trial Evaluating the Safety and Efficacy of GS-6624, a Monoclonal Antibody Against Lysyl Oxidase Like 2 (LOXL2) in Subjects With Primary Sclerosing Cholangitis (PSC)
Brief Title: Simtuzumab (GS-6624) in the Prevention of Progression of Liver Fibrosis in Adults With Primary Sclerosing Cholangitis (PSC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: GS-US-321-0102; 2012-002473-61 (EudraCT Number)
Record Dates: First submitted 2012-08-22; First posted 2012-08-27 (Estimated); Results first posted 2019-10-22 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Primary Sclerosing Cholangitis (PSC)
Keywords: PSC; Sclerosis; Monoclonal antibody; LOXL2; Simtuzumab; Primary sclerosing cholangitis; Liver fibrosis; Liver disease; MRCP; MRE; Liver biopsy
MeSH Terms: conditions — Cholangitis, Sclerosing; Sclerosis; Liver Cirrhosis; Liver Diseases | interventions — simtuzumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment Arm A (Experimental): Simtuzumab 75 mg for 96 weeks
  Interventions: Biological: Simtuzumab
- Treatment Arm B (Experimental): Simtuzumab 125 mg for 96 weeks
  Interventions: Biological: Simtuzumab
- Treatment Arm C (Placebo Comparator): Placebo for 96 weeks
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Simtuzumab — Subcutaneous injections weekly for a total of 96 injections
  Other Names: GS-6624
  Arms: Treatment Arm A; Treatment Arm B
Biological: Placebo — Subcutaneous injections weekly for a total of 96 injections
  Arms: Treatment Arm C

SUMMARY:
The purpose of this study is to evaluate whether simtuzumab (GS-6624) is effective at preventing the progression of liver fibrosis in adults with primary sclerosing cholangitis (PSC).

ELIGIBILITY:
Key Inclusion Criteria:

* Adult Individuals (aged 18-70) with chronic cholestatic liver disease of at least 6 months.
* Liver biopsy consistent with PSC: If a liver biopsy has been performed within 3 months of the screening visit, tissue from that biopsy may be used as the screening biopsy. Slides would be re-cut from the existing tissue block and submitted for central reader assessment. Some individuals with PSC may have a normal liver biopsy, in the event of a normal liver biopsy, the individual must have an abnormal magnetic resonance cholangiopancreatography (MRCP).
* MRCP consistent with PSC: Some individuals with PSC may have a normal MRCP; in the event of a normal MRCP, the individual must have an abnormal liver biopsy.
* Exclusion of other causes of liver disease including viral hepatitis ,alcoholic liver disease,primary biliary cirrhosis and secondary sclerosing cholangitis
* Must have aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 10 x the Central Laboratory Upper Limit of Normal (clULN)
* Must have serum creatinine < 2.0 mg/dL
* A negative serum pregnancy test is required for female individuals of childbearing potential
* All sexually active female individuals of childbearing potential must agree to use a protocol recommended method of contraception during heterosexual intercourse throughout the study and for 90 days following the last dose of study medication
* Lactating females must agree to discontinue nursing before starting study treatment
* Males if not vasectomized, are required to use barrier contraception (condom plus spermicide) during intercourse from the screening through the study completion and for 90 days following the last dose of study drug

Key Exclusion Criteria:

* Pregnant or breast feeding
* Evidence of hepatic decompensation present, including ascites, episodes of hepatic encephalopathy, variceal bleeding or a prolonged prothrombin time/international normalized ratio (PT/INR)
* Positive for hepatitis C virus (HCV) RNA
* Positive for HBsAg
* Positive for anti-mitochondrial antibody
* Alcohol consumption greater than 21oz/week for males or 14oz/week for females
* Moderately active ulcerative colitis (UC) defined as either a partial Mayo score of > 4, bleeding score of >1, or current use of oral corticosteroid therapy and/or any inhibitor of Tumor necrosis factor-α (TNF-α) or α4β7 integrin antagonist
* Positive urine screen for amphetamines, cocaine or opiates (i.e. heroin, morphine) at screening. Individuals on stable methadone or buprenorphine maintenance treatment for at least 6 months prior to screening may be included in the study. Individuals with a positive urine drug screen due to prescription opioid-based medication are eligible if the prescription and diagnosis are reviewed and approved by the investigator
* Clinically significant cardiac disease
* History of cholangiocarcinoma
* History of other cancers,other than non-melanomatous skin cancer, within 5 years prior to screening
* Ascending cholangitis within 60 days of screening
* Presence of a percutaneous drain or bile duct stent
* Known hypersensitivity to the investigation product or any of its formulation excipients
* History of bleeding diathesis within 6 months of screening
* Unavailable for follow-up assessment or concern for individual's compliance with the protocol procedures;
* Participation in an investigational trial of a drug or device within 30 days prior to screening
* Major surgical procedure within 30 days prior to screening or the presence of an open wound

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2013-03-04 (Actual); Primary Completion 2016-08-08 (Actual); Study Completion 2016-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (75):
- United States (43):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - University of Arizona Health Sciences Center, Tucson, Arizona
  - Southern California Liver Center, Chula Vista, California
  - Southern California Liver Centers, Coronado, California
  - Scripps Clinic, La Jolla, California
  - Verterans Adminstration Hospital, Palo Alto, California
  - UC Davis Medical Center, Sacramento, California
  - University of San Diego Medical Center, San Diego, California
  - University of California San Francisco, San Francisco, California
  - University of Colorado Denver, Aurora, Colorado
  - University of Miami Center for Liver Diseases, Miami, Florida
  - Northwestern University, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Indianapolis Gastroenterology Research Foundation, Indianapolis, Indiana
  - Iowa Digestive Disease Center, Clive, Iowa
  - University of Louisville, Louisville, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Minnesota Gastroenterology, PA, Saint Paul, Minnesota
  - St. Louis University, St Louis, Missouri
  - Weill Cornell Medical College, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Duke Clinical Research Institute, Durham, North Carolina
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University Gastroenterology, Providence, Rhode Island
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - St. Luke Episcopal Hospital, Houston, Texas
  - Alamo Medical Research, San Antonio, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Utah, Salt Lake City, Utah
  - University of Virginia Health Center, Charlottesville, Virginia
  - Liver Institute of Virginia, Newport News, Virginia
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - Bon Secours Richmond Health System, Richmond, Virginia
  - Virginia Commonwealth University Health System, Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - University of Washington, Seattle, Washington
- Belgium (5):
  - Hôpital Erasme, Brussels
  - Université Catholique de Louvain, Brussels
  - UZ Antwerpen, Edegem
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
- Canada (6):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - University of Manitoba, Winnepeg, Manitoba
  - Dalhousie University, Halifax, Nova Scotia
  - London Health Science Center, London, Ontario
  - Toronto Liver Centre, Toronto, Ontario
- Denmark (3):
  - Århus Universitetshospital, Århus Sygehus, Århus C
  - Hvidovre Hospital, Hvidovre
  - Rigshospitalet, København Ø
- Germany (4):
  - Klinikum der Johann Wolfgang Goethe Universitat, Frankfurt
  - Medizinische Hochschule Hannover, Hanover
  - Gastroenterologisch Hepatologisches Zentrum Kiel, Kiel
  - EUGASTRO GmbH, Leipzig
- Italy (3):
  - Istituto Clinico Humanitas, Rozzano, Milano
  - Azienda Ospedaliera San Camillo Forlanini, Roma
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino, Torino
- Eramus MC, Rotterdam, Netherlands
- Spain (3):
  - Hospital Universitario Vall d'Hebron, Barcelona, Catalonia
  - Hospital Donostia, Donostia / San Sebastian
  - Hospital Universitario Puerta de Hierro, Majadahonda
- Avd för invärtesmedicin och klinisk nutrition, Gothenburg, Sweden
- United Kingdom (6):
  - New Queen Elizabeth Hospital, Birmingham
  - John Radcliffe Hospital, Headington
  - Imperial College Healthcare NHS Trust- St. Mary's Hospital, London
  - University College London, London
  - Norfolk and Norwich University Hospital, Norwich
  - University of Nottingham, Nottingham

REFERENCES:
- [Result] Shea P, Hirschfield G, Shiffman M, McColgan B, Goodman Z, Myers, R, et al. Common variation near glial-derived neurotrophic factor is associated with progression of hepatic collagen content in a genome-wide association study of liver fibrosis phenotypes in patients with primary sclerosing cholangitis. J Hepatol 2017; 66 (1): S4-S5.
- [Result] Muir A, Goodman Z, Levy C, Janssen H, Montano-Loza A, Bowlus C, et al. Efficacy and safety of simtuzumab for the treatment of primary sclerosing cholangitis: results of a phase 2b, dose-ranging, randomized, placebo-controlled trial. J Hepatol 2017; 66 (1): S73.
- [Result] Bowlus CL, Patel K, Hirschfield G, Guha I, Chapman R, Chazouilleres O, et al. Prospective validation of the Enhanced Liver Fibrosis test for the prediction of disease progression in a randomized trial of patients with primary sclerosing cholangitis. J Hepatol 2017; 66 (1): S359.
- [Result] Levy C, Eksteen B, Shiffman M, Janssen H, Montano-Loza A, Ding D, et al. Prospective validation of serum alkaline phosphatase for the prediction of disease progression in a randomized trial of patients with primary sclerosing cholangitis. J Hepatol 2017; 66 (1): S360-S361.
- [Result] Levy C, Shiffman M, Caldwell S, Luketic V, Invernizzi P, Minuk G, et al. Serum fibroblast growth factor 19, 7α-Hydroxy-4-Cholesten-3-one, and bile acids and their associations with clinical characteristics in primary sclerosing cholangitis. J Hepatol 2017; 66 (1): S361.
- [Result] French D, Huntzicker EG, Goodman ZD, Shea PR, Ding D, Aguilar Schall, RE, et al. Hepatic expression of lysyl oxidase-like-2 (LOXL2) in primary sclerosing cholangitis (PSC). Hepatol 2016; 64 (1): 194A.
- [Result] Bowlus CL, Montano-Loza AJ, Invernizzi P, Chazouilleres O, Hirschfield G, Metselaar HJ, et al. Liver stiffness measurement by transient elastography for the prediction of fibrosis in patients with primary sclerosing cholangitis in a randomized trial of simtuzumab. J Hepatol 2016; 64 (2): S434.
- [Result] Goodman Z, Patel K, Guha I, Hameed B, Kowdley K, Alaparthi L, et al. Correlations between hepatic morphometric collagen content, histologic fibrosis stage, and serum markers in patients with primary sclerosing cholangitis (PSC). J Hepatol 2016; 64 (2): S652-S653.
- [Result] Muir AJ, Goodman Z, Bowlus CL, Caldwell S, Invernizzi P, Luketic V, et al. Serum lysyl oxidase-like-2 (SLOXL2) levels correlate with disease severity in patients with primary sclerosing cholangitis. J Hepatol 2016; 64 (2): S428.
- [Result] Shea PR, Eksteen B, Hirschfield GM, Shiffman ML, Janssen HLA, Montano-Loza AJ, et al. Genome-wide association study (GWAS) of liver fibrosis phenotypes in patients with primary sclerosing cholangitis (PSC) reveals common genetic variation influencing serum levels of lysyl oxidase-like-2 (LOXL2). J Hepatol 2016; 64 (2): S180-S182.
- [Result] Manns MP, Eksteen B, Shiffman ML, Levy C, Kowdley KV, Montano-Loza AJ, et al. Association between elevated serum IgG4 (sIgG4) concentrations and the phenotype of patients with primary sclerosing cholangitis (PSC). Hepatol 2015; 62 (1): 515A.
- [Result] Bowlus CL, Patel K, Chuha IN, Chapman RW, Chazouilleres O, Chalasani NP, et al. Validation of serum fibrosis marker panels in patients with primary sclerosing cholangitis (PSC) in a randomized trial of simtuzumab. Hepatol 2015; 62 (1): 519A.
- [Result] French D, Goodman ZD, Huntzicker EG, Newstrom D, Karnik S, Smith V, et al. Expression of matrix metalloproteinase 9 (MMP9) and the apoptosis signal-regulating kinase 1 (ASK1) pathway activation marker, phospho-P38 (p-P38), in primary sclerosing cholangitis (PSC). Hepatol 2015; 62 (1): 523A-524A.
- [Derived] Laschtowitz A, Lindberg EL, Liebhoff AM, Liebig LA, Casar C, Steinmann S, Guillot A, Xu J, Schwinge D, Trauner M, Lohse AW, Bonn S, Hubner N, Schramm C. Liver transcriptome analysis reveals PSC-attributed gene set associated with fibrosis progression. JHEP Rep. 2024 Nov 12;7(3):101267. doi: 10.1016/j.jhepr.2024.101267. eCollection 2025 Mar. PMID 39996122
- [Derived] Thorburn D, Leeming DJ, Barchuk WT, Wang Y, Lu X, Malkov VA, Ito KL, Bowlus CL, Levy C, Goodman Z, Karsdal MA, Muir AJ, Xu J. Serologic extracellular matrix remodeling markers are related to fibrosis stage and prognosis in a phase 2b trial of simtuzumab in patients with primary sclerosing cholangitis. Hepatol Commun. 2024 Jul 5;8(7):e0467. doi: 10.1097/HC9.0000000000000467. eCollection 2024 Jul 1. PMID 38967589
- [Derived] Muir AJ, Levy C, Janssen HLA, Montano-Loza AJ, Shiffman ML, Caldwell S, Luketic V, Ding D, Jia C, McColgan BJ, McHutchison JG, Mani Subramanian G, Myers RP, Manns M, Chapman R, Afdhal NH, Goodman Z, Eksteen B, Bowlus CL; GS-US-321-0102 Investigators. Simtuzumab for Primary Sclerosing Cholangitis: Phase 2 Study Results With Insights on the Natural History of the Disease. Hepatology. 2019 Feb;69(2):684-698. doi: 10.1002/hep.30237. Epub 2019 Jan 11. PMID 30153359

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in North America and Europe. The first participant was screened on 4 March 2013. The last study visit occurred on 24 August 2016.
Pre-assignment Details: 298 participants were screened.
Groups:
- SIM 75 mg: Simtuzumab (SIM) 75 mg subcutaneous injections weekly for 96 weeks
- SIM 125 mg: SIM 125 mg subcutaneous injections weekly for 96 weeks
- Placebo: Placebo subcutaneous injections weekly for 96 weeks
Period: Overall Study
Arm/Group | SIM 75 mg | SIM 125 mg | Placebo
Started | 79 | 77 | 79
Completed | 69 | 60 | 65
Not Completed | 10 | 17 | 14
Not completed — Protocol Specified Criteria for Withdraw | 0 | 4 | 0
Not completed — Pregnancy | 0 | 1 | 0
Not completed — Investigator's Discretion | 1 | 0 | 0
Not completed — Withdrew Consent | 5 | 5 | 5
Not completed — Adverse Event | 4 | 6 | 8
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Randomized but Never Treated | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included participants who received at least one dose of study drug.
Groups:
- SIM 75 mg: SIM 75 mg subcutaneous injections weekly for 96 weeks
- Total: Total of all reporting groups
Arm/Group | SIM 75 mg | SIM 125 mg | Placebo | Total
Number analyzed (Participants) | 79 | 77 | 78 | 234
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (11.3) | 43 (10.1) | 44 (12.8) | 44 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 25 | 33 | 85
  Male | 52 | 52 | 45 | 149
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 1 | 6
  Not Hispanic or Latino | 78 | 73 | 77 | 228
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 0 | 1 | 3 | 4
  Black | 7 | 6 | 8 | 21
  White | 71 | 68 | 62 | 201
  Other | 1 | 2 | 4 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 16 | 17 | 12 | 45
  Sweden | 1 | 0 | 0 | 1
  Netherlands | 2 | 1 | 2 | 5
  Belgium | 1 | 1 | 1 | 3
  United States | 42 | 35 | 43 | 120
  Denmark | 5 | 3 | 0 | 8
  Italy | 3 | 2 | 5 | 10
  United Kingdom | 5 | 9 | 6 | 20
  Germany | 3 | 2 | 5 | 10
  Spain | 0 | 3 | 2 | 5
  France | 1 | 4 | 2 | 7
Morphometric Quantitative Collagen (MQC) [Mean (Standard Deviation); unit: percentage of MQC] | 5.6 (5.09) | 5.6 (3.36) | 5.1 (3.98) | 5.4 (4.19)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in MQC on Liver Biopsy at Week 96
Time Frame: Baseline; Week 96
Population: Participants in the Full Analysis Set (participants who were randomized into the study and received at least 1 dose of study drug) with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of MQC
Arm/Group | SIM 75 mg | SIM 125 mg | Placebo
Number analyzed (Participants) | 61 | 61 | 62
percentage of MQC | -0.5 (5.78) | 0.5 (6.94) | 0.0 (4.76)
Statistical Analysis 1: Comparison: SIM 75 mg vs Placebo; A mixed-effect model for repeated measures (MMRM) with an unstructured variance-covariance matrix for each participant was used to calculate a point estimate and a 95% confidence interval (CI) for the treatment difference between each treatment arm and placebo in least squares mean (LSMean) change from baseline in MQC at Week 96. With MMRM setting, all participants with available data from the 3 treatment groups with change in MQC at Week 48 and/or Week 96 contributed to the overall model; Test type: Superiority; Difference in LS Mean = -0.4, 95% CI 2-sided [-2.3 to 1.6]
Statistical Analysis 2: Comparison: SIM 125 mg vs Placebo; A MMRM with an unstructured variancecovariance matrix for each participant was used to calculate a point estimate and a 95% CI for the treatment difference between each treatment arm and placebo in LSMean change from baseline in MQC at Week 96. With MMRM setting, all participants with available data from the 3 treatment groups with change in MQC at Week 48 and/or Week 96 contributed to the overall model; Test type: Superiority; Difference in LS Mean = 1.0, 95% CI 2-sided [-1.0 to 3.0]

2. Secondary Outcome: Percentage of Participants Who Permanently Discontinued Any Study Drug Due to an Adverse Event
Time Frame: First dose date up to Week 96
Population: The Safety Analysis Set included participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | SIM 75 mg | SIM 125 mg | Placebo
Number analyzed (Participants) | 79 | 77 | 78
percentage of participants | 5.1 | 7.8 | 10.3

3. Secondary Outcome: Study Drug Exposure
Description: The average SIM exposure was summarized.
Time Frame: First dose date up to Week 96
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | SIM 75 mg | SIM 125 mg | Placebo
Number analyzed (Participants) | 79 | 77 | 78
weeks | 92.0 (15.33) | 83.8 (26.12) | 87.4 (22.35)

4. Secondary Outcome: Percentage of Participants Experiencing Any Treatment-Emergent Laboratory Abnormality
Description: A treatment-emergent graded laboratory abnormality was defined as an increase of at least 1 abnormality grade from the predose assessment and occurring after the predose visit and on or before the date of the administration of study drug plus 30 days. The most severe graded abnormality from all tests was counted for each participant [Grade 1 (mild); Grade 2 (moderate); Grade 3 (severe); Grade 4 (life-threatening)].
Time Frame: First dose date up to Week 96 plus 30 days
Population: Participants in the Safety Analysis Set with at least one post-baseline measurement were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | SIM 75 mg | SIM 125 mg | Placebo
Number analyzed (Participants) | 79 | 77 | 78
percentage of participants
  Grade 1 | 11.4 | 16.9 | 17.9
  Grade 2 | 26.6 | 20.8 | 25.6
  Grade 3 | 48.1 | 46.8 | 48.7
  Grade 4 | 11.4 | 13.0 | 7.7

ADVERSE EVENTS:
Time Frame: First dose date up to Week 96 plus 30 days
Description: The Safety Analysis Set included participants who received at least one dose of study drug.
Arm/Group | SIM 75 mg | SIM 125 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/79 | 0/77 | 0/78
Serious Adverse Events (participants affected / at risk) | 16/79 | 23/77 | 21/78
Other Adverse Events (participants affected / at risk) | 71/79 | 72/77 | 75/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SIM 75 mg (N=79) | SIM 125 mg (N=77) | Placebo (N=78)
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 3 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1 | 0
Diverticular perforation (Gastrointestinal disorders) | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 1
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 1 | 1
Cholangitis (Hepatobiliary disorders) | 6 | 5 | 3
Cholangitis acute (Hepatobiliary disorders) | 0 | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 1 | 1
Gallbladder perforation (Hepatobiliary disorders) | 1 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 1
Cholangitis infective (Infections and infestations) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 1 | 0
Infected skin ulcer (Infections and infestations) | 0 | 1 | 0
Pelvic abscess (Infections and infestations) | 0 | 0 | 1
Peritonitis (Infections and infestations) | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 2
Sepsis (Infections and infestations) | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 0 | 1
Streptococcal bacteraemia (Infections and infestations) | 1 | 0 | 0
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Postoperative fever (Injury, poisoning and procedural complications) | 0 | 1 | 1
Procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 1
Stoma obstruction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0
Liver function test increased (Investigations) | 0 | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Benign biliary neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1
Post-traumatic stress disorder (Psychiatric disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SIM 75 mg (N=79) | SIM 125 mg (N=77) | Placebo (N=78)
Anaemia (Blood and lymphatic system disorders) | 4 | 3 | 4
Abdominal discomfort (Gastrointestinal disorders) | 4 | 4 | 3
Abdominal distension (Gastrointestinal disorders) | 4 | 3 | 6
Abdominal pain (Gastrointestinal disorders) | 13 | 18 | 17
Abdominal pain lower (Gastrointestinal disorders) | 2 | 3 | 4
Abdominal pain upper (Gastrointestinal disorders) | 18 | 14 | 18
Colitis ulcerative (Gastrointestinal disorders) | 1 | 1 | 5
Constipation (Gastrointestinal disorders) | 7 | 1 | 7
Diarrhoea (Gastrointestinal disorders) | 19 | 15 | 15
Dyspepsia (Gastrointestinal disorders) | 2 | 2 | 9
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 5
Haemorrhoids (Gastrointestinal disorders) | 4 | 1 | 0
Nausea (Gastrointestinal disorders) | 16 | 17 | 17
Rectal haemorrhage (Gastrointestinal disorders) | 5 | 2 | 3
Varices oesophageal (Gastrointestinal disorders) | 2 | 5 | 4
Vomiting (Gastrointestinal disorders) | 9 | 5 | 7
Asthenia (General disorders) | 1 | 4 | 3
Fatigue (General disorders) | 19 | 21 | 16
Influenza like illness (General disorders) | 3 | 4 | 4
Injection site erythema (General disorders) | 2 | 5 | 0
Injection site pain (General disorders) | 4 | 0 | 3
Pain (General disorders) | 0 | 6 | 5
Pyrexia (General disorders) | 11 | 10 | 13
Cholangitis (Hepatobiliary disorders) | 6 | 6 | 4
Jaundice (Hepatobiliary disorders) | 5 | 4 | 3
Bronchitis (Infections and infestations) | 2 | 3 | 7
Gastroenteritis (Infections and infestations) | 2 | 5 | 2
Gastroenteritis viral (Infections and infestations) | 5 | 1 | 4
Influenza (Infections and infestations) | 5 | 2 | 7
Lower respiratory tract infection (Infections and infestations) | 5 | 0 | 1
Nasopharyngitis (Infections and infestations) | 19 | 17 | 14
Sinusitis (Infections and infestations) | 5 | 11 | 5
Upper respiratory tract infection (Infections and infestations) | 11 | 9 | 10
Urinary tract infection (Infections and infestations) | 6 | 4 | 4
Contusion (Injury, poisoning and procedural complications) | 4 | 3 | 0
Procedural pain (Injury, poisoning and procedural complications) | 4 | 7 | 7
Blood bilirubin increased (Investigations) | 4 | 2 | 3
Decreased appetite (Metabolism and nutrition disorders) | 4 | 3 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 12 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 8 | 9
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 2 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 3 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 7 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 2 | 4
Dizziness (Nervous system disorders) | 6 | 5 | 4
Headache (Nervous system disorders) | 18 | 12 | 17
Anxiety (Psychiatric disorders) | 2 | 3 | 4
Insomnia (Psychiatric disorders) | 5 | 5 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 7 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 4
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 21 | 22 | 31
Rash (Skin and subcutaneous tissue disorders) | 10 | 2 | 3
Hypertension (Vascular disorders) | 3 | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years